CLINICAL TRIAL: NCT00242931
Title: Pilot Trial of Non-Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation for the Treatment of Patients With Hormone-Refractory Prostate Cancer
Brief Title: Flu/TBI in Treating Patients Not Responding to Previous Hormone Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to successfully recruit subjects to this study.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000447211; OHSU-SOL-04109-L (Other: OHSU); OHSU-373 (Other: OHSU)
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2010-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fludarabine, TBI, Cyclosporine, MMF (Experimental): Fludarabine 30 mg/m2/day x 3, day -4 to day -2 TBI 200 cGy x 1, day 0 For related donors: cyclosporine (CSP) 5 mg/kg p.o. bid, day -3 to day +56, then taper by 20% every 5 days to be completed by day +81 For related donors: mycophenolate mofetil (MMF) 15 mg/kg p.o. q 12 hours, day 0 to day +27, then stop
  For unrelated donors: cyclosporine (CSP) 5 mg/kg p.o. bid, day -3 to day +56, then taper by 20% every 5 days to be completed by day +81 For unrelated donors: mycophenolate mofetil (MMF) 15 mg/kg tid day +0 to day +29, 15 mg/kg bid day +30 to day +149, and then taper by 25% per week from day +150 to day +180. Discontinue by day +181.
  Interventions: Other: Nonmyeloablative stem cell conditioning regimen

INTERVENTIONS:
Other: Nonmyeloablative stem cell conditioning regimen — Conditioning:
  Fludarabine 30 mg/m2/day x 3, day -4 to day -2 TBI 200 cGy x 1, day 0
  Hematopoeitic Stem Cell Transplantation:
  Infusion of peripheral blood stem cells, day 0
  Immunosuppression:
  For related donors: cyclosporine (CSP) 5 mg/kg p.o. bid, day -3 to day +56, then taper by 20% every 5 days to be completed by day +81 For related donors: mycophenolate mofetil (MMF) 15 mg/kg p.o. q 12 hours, day 0 to day +27, then stop
  For unrelated donors: cyclosporine (CSP) 5 mg/kg p.o. bid, day -3 to day +56, then taper by 20% every 5 days to be completed by day +81 For unrelated donors: mycophenolate mofetil (MMF) 15 mg/kg tid day +0 to day +29, 15 mg/kg bid day +30 to day +149, and then taper by 25% per week from day +150 to day +180. Discontinue by day +181.
  Other Names: Mini Transplant

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine, and radiation therapy before a donor stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving fludarabine together with total-body irradiation works in treating patients who are undergoing a donor stem cell transplant for progressive metastatic prostate cancer that has not responded to previous hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the treatment-related mortality in patients with hormone-refractory, progressive metastatic prostate cancer treated with nonmyeloablative conditioning comprising fludarabine and total-body irradiation followed by allogeneic hematopoietic stem cell transplantation.

OUTLINE:

* Nonmyeloablative conditioning regimen: Patients receive fludarabine IV on days -4 to -2 and total-body irradiation (TBI) on day 0.
* Allogeneic hematopoietic stem cell transplantation (AHSCT): After TBI, patients undergo AHSCT on day 0.
* Immunosuppression: Patients receive oral cyclosporine twice daily on days -3 to 56 followed by a taper until day 81. Patients also receive oral mycophenolate mofetil twice daily on days 0-27 (if patient has a related donor) OR three times daily on days 0-29 and then twice daily on days 30-149 followed by additional tapering until day 180 (if patient has an unrelated donor).

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adenocarcinoma of the prostate

  * Metastatic and progressive disease
  * Refractory to hormonal therapy
* Prostate-specific antigen (PSA) > 5 ng/mL
* Previously treated with a docetaxel-based regimen
* No CNS metastases

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 70-100%

Life expectancy

* More than 6 months

Hematopoietic

* Not specified

Hepatic

* Bilirubin < 2 times upper limit of normal (ULN)
* AST and ALT < 4 times ULN

Renal

* Creatinine clearance > 50 mL/min

Cardiovascular

* LVEF > 35%
* No symptomatic congestive heart failure

Pulmonary

* DLCO > 40% of predicted OR
* Total lung capacity or FEV_1 > 30% of predicted

Other

* HIV negative

PRIOR CONCURRENT THERAPY:

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* See Disease Characteristics

PATIENT AND DONOR SELECTION CRITERIA

4.1 Patient Inclusion Criteria:

4.1.1 Males aged 18-75.

4.1.2 Pathologically proven adenocarcinoma of the prostate with metastases and progressive disease (new metastatic lesions or increase in cancer-related pain or a rising PSA defined by consensus criteria. (A rising PSA will be defined as 2 measurements higher than an initial value. The second of the 3 measurements must be at least 7 days after the first).

4.1.3 Progressive disease despite hormonal management (including antiandrogen withdrawal, 6 weeks for bicalutamide, 4 weeks for flutamide or nilutamide)

4.1.4 PSA > 5 ng/mL

4.1.5 Serum testosterone level < 50 ng/mL

4.1.6 Prior treatment with a docetaxel-based regimen.

4.1.7 Performance status: Karnofsky Performance Scale (KPS) 70-100%. (Appendix III).

4.1.8 Signed informed patient consent.

4.2 Patient Exclusion criteria:

4.2.1 Expected survival less than 6 months

4.2.2 Active central nervous system involvement or spinal instability

4.2.3 Organ dysfunction:

4.2.3.1 Cardiac: Ejection fraction <35% or symptomatic congestive heart failure.

4.2.3.2 Pulmonary: DLCO <40% of predicted or either TLC or FEV1 < 30% predicted.

4.2.3.3 Liver dysfunction: serum total bilirubin >2x upper limit of normal (ULN) or either ALT or AST >4x ULN

4.2.3.4 Renal dysfunction: creatinine clearance < 50 ml/min

4.2.4 HIV seropositivity

4.2 Related Donor Inclusion criteria:

4.3.1 Age 18-75

4.3.2 Related to the patient and genotypically or phenotypically HLA-identical. (Appendix IV)

4.3.3 Able to give consent to peripheral blood stem cell mobilization with G-CSF and apheresis collection. Bone marrow donors are not eligible.

4.3 Unrelated Donor Inclusion criteria:

4.4.1 Age 18-75.

4.4.2 Unrelated donors who are prospectively:

4.4.2.1 Matched for HLA-DRB1 and -DQB1 alleles by high resolution typing AND 4.4.2.2 Matched for all serologically recognized HLA-A or -B or -C antigens and at least five of six HLA-A or -B or -C alleles as defined by Appendix IV.

4.4.3 Able to give consent to peripheral blood stem cell mobilization with G-CSF and apheresis collection. Bone marrow unrelated donors are not eligible.

4.4 Related and Unrelated Donor Exclusion criteria:

4.5.1 Identical twin.

4.5.2 Any contraindication to the administration of G-CSF for mobilization.

4.5.3 Serious medical or psychological illness.

4.5.4 Prior malignancy within the preceding five years, with the exception of non-melanoma skin cancers.

4.5.5 HIV seropositivity.

4.5.6 The donor is pregnant, has a positive serum ßhCG or is lactating.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Treatment-related mortality as measured by Kaplan-Meier at 5 years following transplant

SECONDARY OUTCOMES:
Safety by CTCAE v 3.0 at 100 days following transplant
Response rate by RECIST criteria at 5 years following transplant
Time to progression by Kaplan-Meier at 5 years following transplant
Overall survival by Kaplan-Meier at 5 years following transplant
Response as measured by a 50% reduction in the prostate-specific antigen at 5 years following transplant

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M. Hayes-Lattin, MD, Study Chair — Oregon Health and Science University